CLINICAL TRIAL: NCT04409600
Title: Comparison of Non-Surgical Treatment Options for Chronic Exertional Compartment Syndrome (CECS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: WRNMMC-2019-0266
Record Dates: First submitted 2020-05-07; First posted 2020-06-01 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Exertional Compartment Syndrome
Keywords: botulinum toxin, gait training, military
MeSH Terms: conditions — Chronic Exertional Compartment Syndrome | interventions — Sodium Chloride; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are masked to treatment injection arm. At 3 months post-injection, the treatment injection arm will be revealed to the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Home Based Gait Retraining + Saline Injection (Active Comparator)
  Interventions: Behavioral: Home Based Gait Retraining; Drug: Saline Injection
- Home Based Gait Retraining + Botulinum Toxin Injection (Experimental)
  Interventions: Behavioral: Home Based Gait Retraining; Drug: Botulinum Toxin Injection
- Supervised Gait Retraining + Saline Injection (Active Comparator)
  Interventions: Behavioral: Supervised Gait Retraining; Drug: Saline Injection
- Supervised Gait Retraining + Botulinum Toxin Injection (Experimental)
  Interventions: Behavioral: Supervised Gait Retraining; Drug: Botulinum Toxin Injection

INTERVENTIONS:
Behavioral: Supervised Gait Retraining — The participants allocated to this group will attend 8 sessions during the course of 6 weeks in the clinic with a trained medical professional to complete a supervised gait retraining program.
  Arms: Supervised Gait Retraining + Botulinum Toxin Injection; Supervised Gait Retraining + Saline Injection
Behavioral: Home Based Gait Retraining — The participants allocated to this group will have 1 session in the clinic with a trained medical professional and be given a gait retraining program to complete at home.
  Arms: Home Based Gait Retraining + Botulinum Toxin Injection; Home Based Gait Retraining + Saline Injection
Drug: Saline Injection — The participant will receive a saline injection to their painful lower leg compartment(s).
  Arms: Home Based Gait Retraining + Saline Injection; Supervised Gait Retraining + Saline Injection
Drug: Botulinum Toxin Injection — The participant will receive a botulinum toxin injection to their painful lower leg compartment(s).
  Arms: Home Based Gait Retraining + Botulinum Toxin Injection; Supervised Gait Retraining + Botulinum Toxin Injection

SUMMARY:
Chronic Exertional Compartment Syndrome (CECS) in the lower leg is a debilitating condition in highly active individuals. Pain occurs in 1 or several leg compartments upon an exertional activity, typically running, that quickly dissipates once the activity stopped. Surgical fasciotomy is the standard for treating lower leg CECS, but success is variable. Complications may occur post-surgery and there is a potential for a repeat procedure. Recovery times post-surgery also vary greatly. Conservative treatments, such as gait retraining and botulinum toxin injections, are emerging as non-surgical options for the treatment of CECS with success through published case reports and case series. This study aims to evaluate the use of these non-surgical treatment options for CECS in the anterior and lateral leg compartments with a follow up for at least 2 years across multiple study sites.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service
* Fluent in speaking and reading English
* Unable to run 2 miles without producing pain and/or symptoms
* Difficulty completing the running portion of their service-specific physical training due to pain and/or symptoms in their lower leg
* Meets clinical diagnostic criteria for CECS of the anterior or lateral compartment per clinical examination (palpation, intramuscular compartment pressure, lower leg MRI).

Exclusion Criteria:

* Prior botulinum injection in the lower leg compartment of the affected limb
* Prior compartment release of affected lower leg
* Recent (within the last 6 months) lower limb injury that needed medical intervention
* Completed formal gait retraining within the last 6 months
* Allergic to botulinum toxin
* Pregnant or breastfeeding
* Medical examination that indicates a condition other than CECS

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Balance Error Scoring System Score | baseline, 6 weeks, 3-, 6-, 12-months post injection
  Clinical evaluation tool to assess balance. Individuals are assessed on a firm and flat surface while completing different stances and observed for multiple errors while performing the activity. The higher the number of errors, the greater the deficiency in their balance.
Change in University of Wisconsin Running Injury and Recovery Index Score | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  9-item questionnaire that assesses an individual's ability to run after a running related injury. Total maximum score is 36 with higher scores indicating no deficiency in their ability to run.
Change in Single Assessment Numerical Evaluation (SANE) | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  A patient reported outcome measure consisting of 1 question that asks the individual to rate their current level of function compared to their function prior to their injury, on a scale from 0-100. A higher score suggests a higher level of function.
Change in Patient Specific Functional Scale Scores | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Individuals are asked to self-assess limited activities and measure them on a scale from 0-10 where '0' indicates they are able to perform the activity and '10' indicates that they are unable to perform the activity prior to their condition.
Change in Global Rate of Change Score | 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Using a 15 point scale, the individual selects 1 choice to reflect their current perceived health rating compared to a specified time point.
Change in gait analysis | baseline, 6 weeks, 3-, 6-, 12-months post injection
  Using wearable technology and slow motion capture camera, gait analysis will be collected.
Change in ability to return to full active duty | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Question asked to military service members about their ability to return to full active duty.
Change in ability to run 2 miles | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Question asked to military service members about their ability to run 2 miles.

SECONDARY OUTCOMES:
Pain reduction | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Pain reduction will be assessed using a numeric pain rating scale (NPRS). This is an 11 point Likert scale that reflects the individual's pain level.
Ability to perform service specific military physical training requirements | baseline, 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Question that asks the military service member of their ability to perform service specific physical training requirements.
Patient satisfaction of treatment | 6 weeks, 3-, 6-, 12-, 24-, 36-months post injection
  Questionnaire asking the individual to rate their satisfaction of treatment from 'exceptional' to 'very poor.'

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Leggit, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (4):
- United States (4):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Carl R. Darnell Army Medical Center, Killeen, Texas
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

DOCUMENTS (1):
  • Informed Consent Form (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04409600/ICF_000.pdf